CLINICAL TRIAL: NCT04608890
Title: Eye-tracking-based Artificial Intelligence Detects Abnormalities of the Oculomotor System in Type 1 Diabetes
Acronym: EyekonT1D
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Collaborators: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Associate Professor of Endocrinology, University of Milan
Other Study IDs: EyekonT1D
Record Dates: First submitted 2020-10-08; First posted 2020-10-29 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long-standing T1D patients: Patients with long-standing type 1 diabetes
  Interventions: Diagnostic Test: Eye-tracking video test
- Healthy volunteers: Healthy volunteers
  Interventions: Diagnostic Test: Eye-tracking video test

INTERVENTIONS:
Diagnostic Test: Eye-tracking video test — An eye-tracking-based test will be administered to patients. It lasts 10 minutes. It consists in several screens passing by to identify objects at a certain time by a mouse clic or touchpad.

SUMMARY:
Abnormalities of the oculomotor system may represent an early sign of diabetic neuropathy and are currently poorly studied. The investigators designed an eye-tracking-based test to evaluate the oculomotor function in patients with type 1 diabetes.

The investigators used the SRLab -Tobii TX300 Eye tracker®, an eye-tracking device, coupled with a software that we developed to test abnormalities of the oculomotor system. The software consists in a series of screens divided in 5 classes of parameters (Resistance, Wideness, Pursuit, Velocity and Optokinetic Nystagmus [OKN]) to evaluate both smooth and saccadic movement in different directions. 40 healthy volunteers and 40 patients with long-standing type 1 diabetes will be enrolled to analyze the alterations in the oculomotor system and function.

DETAILED DESCRIPTION:
The study will enroll 40 healthy volunteers and 40 patients with long-standing type 1 diabetes. The aim of the study is to analyze alterations in the oculomotor system function as an early sign of diabetic neuropathy. A novel eye-tracking-based test will be employed and 5 parameters will be analyzed through the use of a computer-based test which will record timeframes of eye movements towards an object, type of eye movements, time between the first eye movement, number of visualization required to recognize the object across the screen. Each of these parameter will be employed to assess whether Resistance, Wideness, Pursuit, Velocity of eye movements and movements related to the Optokinetic Nystagmus are altered in type 1 diabetes as compared to non diabetic subjects.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Type 1 diabetes
* willing to give consent

Exclusion Criteria:

* Diabetic retinopathy and other ocular diseases
* other endocrine disease
* malignancy

Healthy volunteers:

Inclusion Criteria:

* willing to give consent

Exclusion Criteria:

* Other ocular diseases
* Any endocrine disease
* Malignancy

Ages: 16 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: N=40 patients with type 1 diabetes on insulin treatment N=40 healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a change in eye movement test in each class Resistance, Velocity, Pursuit, Wideness and OKN measured by the eye-tracking based test | End of the study (when all patients have completed all sessions of the test), an average of 6 months
  Percentage of all parameters tested in each class changed in patients with type 1 diabetes as compared to healthy subjects. Parameters evaluated include number of visualization required to recognize a target and time (seconds), to recognize a target moving on the screen in different directions.

SECONDARY OUTCOMES:
Percentage of patients with a change in eye movement test in the Resistance class | End of the study (when all patients have completed all sessions of the test), an average of 6 months
  Percentage of parameters tested in the Resistance class changed in patients with type 1 diabetes as compared to healthy subjects. Resistance will be measured by using number of visualization required to recognize a target and time (seconds) required to recognize a target moving on the screen in different directions. An algorithm will attribute those measurements to the specific class of Resistance.
Percentage of patients with a change in eye movement test in the Wideness class | End of the study (when all patients have completed all sessions of the test), an average of 6 months
  Percentage of parameters tested in the Wideness class changed in patients with type 1 diabetes as compared to healthy subjects. Wideness will be measured by using number of visualization required to recognize a target and time (seconds) required to recognize a target moving on the screen in different directions. An algorithm will attribute those measurements to the specific class of Wideness.
Percentage of patients with a change in eye movement test in the Velocity class | End of the study (when all patients have completed all sessions of the test), an average of 6 months
  Percentage of parameters tested in the Velocity class changed in patients with type 1 diabetes as compared to healthy subjects. Velocity will be measured by using number of visualization required to recognize a target and time (seconds) required to recognize a target moving on the screen in different directions. An algorithm will attribute those measurements to the specific class of Velocity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sacco University Hospital, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be shared under MTA agreement.

REFERENCES:
- [Derived] D'Addio F, Pastore I, Loretelli C, Valderrama-Vasquez A, Usuelli V, Assi E, Mameli C, Macedoni M, Maestroni A, Rossi A, Lunati ME, Morpurgo PS, Gandolfi A, Montefusco L, Bolla AM, Ben Nasr M, Di Maggio S, Melzi L, Staurenghi G, Secchi A, Bianchi Marzoli S, Zuccotti G, Fiorina P. Abnormalities of the oculomotor function in type 1 diabetes and diabetic neuropathy. Acta Diabetol. 2022 Sep;59(9):1157-1167. doi: 10.1007/s00592-022-01911-1. Epub 2022 Jun 22. PMID 35729357